CLINICAL TRIAL: NCT04441762
Title: Atomized Intranasal Vs Intravenous Ketorolac in Acute Renal Colic Pain Management: A Randomized Controlled Double-blinded Clinical Trial.
Brief Title: Atomized Intranasal Vs Intravenous Ketorolac in Acute Renal Colic Pain Management.
Acronym: Ink-Arc
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Usama Al-Khalasi, Emergency Medicine Resident, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InkArc2020
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: case-control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous (Active Comparator): 30 mg intravenous ketorolac in 10 ml syringe + 1 mL Normal Saline 9% using an intranasal device (0.5 ml in each nostril).
  Interventions: Drug: Intravenous Ketorolac Tromethamine
- Intranasal (Experimental): 30 mg intranasal ketorolac in 1 ml intranasal device (0.5 ml in each nostril) + 10 ml Intravenous Normal Saline 9%.
  Interventions: Drug: Intranasal Ketorolac Tromethamine

INTERVENTIONS:
Drug: Intravenous Ketorolac Tromethamine — 30 mg ketorolac single dose
  Other Names: ketorolac injection
  Arms: intravenous
Drug: Intranasal Ketorolac Tromethamine — 30 mg ketorolac single dose
  Other Names: Atomized Intranasal Ketorolac
  Arms: Intranasal

SUMMARY:
Introduction: Pain is a common reason for individuals to seek health care, especially emergency care. Ketorolac has numerous advantages over other pain medications, especially the opioids. The intranasal administration of ketorolac has been shown to be safe and effective in the treatment of postoperative pain following major abdominal surgery and post dental surgery, but there have been no studies evaluating the use of intranasal ketorolac for the treatment of acute renal colic pain in the emergency department.

Methods: This is a double blinded randomized controlled trial. two hundred renal colic patients presented to the emergency department will be randomized to intervention (30 mg intranasal ketorolac) and (30mg intravenous ketorolac) case groups. Their pain before and after receiving ketorolac will be measured by visual Analog Scale (VAS pain score). Patient, attending physician and administering nurse will be blinded throughout the study. The analgesic effects will be assessed by several measures including pain relief, pain intensity difference, global pain evaluation, global assessment of analgesia, and the summed pain intensity difference. The safety will be assessed by documentation of adverse events, vital signs, and clinical assessment before and after drug administration.

Aim: The aim of this study is to compare analgesic effects of intranasal Ketorolac tromethamine versus intravenous Ketorolac tromethamine in adult patients with moderate to severe renal colic.

Primary Objective: Analgesic effects of Intranasal Ketorolac on the visual analog scale (VAS).

Secondary Objectives: Adverse Events, the need of rescue pain medications, time to discharge and recurrent visit within 24 hours.

Patient Population: Adults (from age 18 to 64 years) who presents to emergency department (ED) at Sultan Qaboos University Hospital with moderate to severe acute flank pain suggestive of renal colic (visual analog scale 7 or more).

Intervention: Single dose of intranasal ketorolac 30mg.

Clinical measurement: Visual Analog Scale will be assessed at 0, 30 and 60 minutes after intervention. Number and dosage of rescue medication, any reported events by patient or attending physician will be documented.

Outcome: Decrease in pain measures by VAS pain score after intranasal ketorolac is given, tolerability and safety evaluation.

DETAILED DESCRIPTION:
Research objectives and hypothesis:

The aim of this study is to compare the analgesic effects of intranasal Ketorolac tromethamine versus intravenous Ketorolac tromethamine in adult patients with moderate to severe renal colic seen at the Emergency Department at Sultan Qaboos University Hospital.

Study design:

Prospective double-blinded randomized clinical trial in adults (from age 18 to 64 years) who presents to the emergency department (ED) at Sultan Qaboos University Hospital with moderate to severe acute flank pain suggestive of renal colic (visual analog scale 7 or more). Written consent will be obtained from the patient. Eligible subjects will be enrolled (see section 5).

Control Group Will receive 30 mg intravenous ketorolac in 10 ml syringe + 1 ml Normal Saline 9% using the intranasal device (0.5 ml in each nostril).

Intervention Group Will receive 30 mg intranasal ketorolac in 1 ml intranasal device (0.5 ml in each nostril) + 10 ml Intravenous Normal Saline 9%.

Primary endpoint:

Analgesic effects of Intranasal Ketorolac on the visual analog scale (VAS). Change in visual analog scale after receiving intranasal ketorolac. 0 (no pain) - 10 (worst possible pain).

Secondary endpoint:

* Adverse Event/Side Effects.
* Safety assessed by reporting all adverse events.
* The need of rescue pain medications.
* Time to discharge.
* Recurrent visit within 24 hours.

Sample size:

after 1 hour follow-up, 146 patient will be needed ( 73 on each arm) to have 90% power to detect a difference of a 0.7 of the response of visual analog scale score ( which usually ranges between 0 and 10 ) between the groups (5.3 vs 4.6) at the 5% alpha (significance) level. Because of missing data and losses to follow-up, an additional 54 subjects will be needed (100 in each arm) for a total of 200 subjects (study sample). A P-value <0.5. Level of significance to be used.

Study Procedures:

1. Present to the Clinical Site Adult subjects ages 18 to 64 years with a classical presentation of acute renal colic being seen in the emergency department may be eligible for this study.

   Clinical sign and symptoms
   * Severe flank pain radiating inferiorly and anteriorly with or without:
   * Nausea and vomiting.
   * Urinary symptoms.
   * Previous history of renal colic.
2. Eligibility Assessments Inclusion and exclusion criteria will be check.
3. Informed Consent Potentially eligible participants will be identified by their treating clinicians. Written informed consent to participate in this study will follow a process of information exchange between clinicians and potential participants.
4. Study Pain Assessments

   Three pain assessments will be done based on VAS-Pain at:
   * 0 minutes
   * 30 minutes
   * 60 minutes Pain scores will be recorded and documented before the administration of medication for a baseline pain assessment and at specified intervals after the administration. Post-treatment pain scores will be recorded at 0, 30 and 60 minutes. Pain assessments will be by the Visual Analog Scale for Pain. It is usually presented as a 10cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." All patients must have a minimum of two pain scores. If rescue medications were given, a VAS-Pain will be obtained immediately prior to treatment.
5. Standard-of-Care Procedures: Pain Management Patients may receive additional medications as part of their emergency department treatment including additional pain medications, such as opioids. Any additional medications administered will be recorded. The need for additional medications (including the drug administered, the dose, the time, and the route of administration) will be recorded.
6. Safety Assessments All adverse events will be documented on an adverse event case log. Serious adverse events should be immediately reported to the primary investigator. Any serious, adverse event will be reported immediately to the Institutional Review Board.

Adverse Events is considered serious if it causes a threat to the patient's life or functioning. The U.S. Food and Drug Administration (FDA) defines a serious adverse event (SAE) as any untoward medical occurrence that:

* Results in death.
* Life-threatening (places the patient at risk of death).
* Requires hospitalization or prolongs an existing hospitalization.
* Causes persistent or significant disability or incapacity.
* Requires medical intervention to prevent one of the above outcomes.

RISKS AND BENEFITS Ketorolac has been proven effective for pain relief, especially for certain types of pain, such as musculoskeletal pain, headaches and the pain from renal colic. Inappropriate patients, ketorolac is a relatively safe drug for the treatment of pain. Side effects and complications, such as gastrointestinal complaints (e.g. abdominal pain, dyspepsia, GI bleeding) and renal dysfunction (elevation of the blood urea nitrogen and creatinine) have been reported but with appropriate patient's selection are uncommon or rare. The use of NSAIDS including ketorolac is not recommended in patients with active peptic ulcer disease, renal disease or at risk for renal failure due to volume depletion, cerebrovascular bleeding, hemorrhagic disorders, or those with a high risk of bleeding. With an appropriate patient selection, ketorolac can be a safe and effective medication for the relief of pain. The drug used in this study has a very low risk of developing any complications. However, during visits patients will be monitored for any complications and all adverse effects if any will be reported. With the proposed hypothesis, intranasal has the potential to reduce opioid use in the ED, provides fast, needleless and easy methods to apply. It will decrease the waiting time, cannulation and unnecessary blood investigations in patients with a classic presentation of acute renal colic.

ELIGIBILITY:
Inclusion Criteria:

* Patient with classical acute renal colic symptoms.
* Age ≥ 18 years and < 65 years
* Stable patient with stable vital signs.
* Mentally competent patient who can understand and sign the consent form.
* Pain score is moderate to severe (visual analog scale 7 or more).

Exclusion Criteria:

* Patients who are allergic to ketorolac.
* Patients with active peptic ulcer disease.
* Patients with a history of asthma, urticaria, or other allergic-type reactions after taking NSAIDs.
* Patients with renal disease and renal transplant.
* Patients who are at risk for renal failure due to volume depletion.
* Pregnant or nursing mothers.
* Patients with any other contraindication to the use of ketorolac, or in whom the use of ketorolac would not be consistent with the approved package insert.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Analgesic effects of Intranasal Ketorolac on the visual analog scale (VAS) | At 30 and 60 minutes
  Change in visual analog scale after receiving intranasal ketorolac. 0 (no pain) - 10 (worst possible pain).

SECONDARY OUTCOMES:
Adverse Events/Side Effects. | 48 hours
  Any reported adverse events reported by subjects or attending doctor
The need of rescue pain medications. | 60 min During Emergency Visit
  After 60 min , patients can have rescue medications as standard of care.
Time to discharge. | within 24 hours.
  The time since first dose of Ketorolac to ED discharge.
Recurrent visit | within 24 hours.
  Any recurrent visit with acute renal colic complaint

CONTACTS AND LOCATIONS:
Overall Officials: Usama Al-Khalasi, Principal Investigator — Oman Medical Speciality Board
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Aseeb, Oman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arhami Dolatabadi A, Memary E, Kariman H, Nasiri Gigloo K, Baratloo A. Intranasal Desmopressin Compared with Intravenous Ketorolac for Pain Management of Patients with Renal Colic Referring to the Emergency Department: A Randomized Clinical Trial. Anesth Pain Med. 2017 Feb 25;7(2):e43595. doi: 10.5812/aapm.43595. eCollection 2017 Apr. PMID 28824859
- [Result] Yazdani J, Khorshidi-Khiavi R, Nezafati S, Mortazavi A, Farhadi F, Nojan F, Ghanizadeh M. Comparison of analgesic effects of intravenous and intranasal ketorolac in patients with mandibular fracture-A Randomized Clinical Trial. J Clin Exp Dent. 2019 Sep 1;11(9):e768-e775. doi: 10.4317/jced.55753. eCollection 2019 Sep. PMID 31636867
- [Result] Singla N, Singla S, Minkowitz HS, Moodie J, Brown C. Intranasal ketorolac for acute postoperative pain. Curr Med Res Opin. 2010 Aug;26(8):1915-23. doi: 10.1185/03007995.2010.495564. PMID 20557145